CLINICAL TRIAL: NCT00778401
Title: A Relative Bioavailability Study of 800 mg Gabapentin Tablets Under Fasting Condition
Brief Title: Bioequivalence Study of Gabapentin 800 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R01-825
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Gabapentin tablets 800 mg fasting conditions
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Gabapentin tablets 800 mg by Ranbaxy Laboratories Limited
  Interventions: Drug: Gabapentin tablets 800 mg
- 2 (Active Comparator): Neurontin ® 800 mg tablets of Parke Davis Pharmaceuticals Ltd.
  Interventions: Drug: Gabapentin tablets 800 mg

INTERVENTIONS:
Drug: Gabapentin tablets 800 mg

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of the test Gabapentin tablets 800 mg by Ranbaxy Laboratories Limited to the reference Neurontin ® 800 mg tablets of Parke Davis Pharmaceuticals Ltd., distributed by Parke Davis, division of Warner-Lambert Co. in 28 healthy, adult subjects (21 males and 7 females) under fasting conditions using randomized, two-way crossover design.

DETAILED DESCRIPTION:
A single oral dose of the test or reference product was administered to the volunteers on two separate occasions under fasting conditions with at least a 7 day washout between doses. Food and fluid intake were controlled during each confinement period.

A total of twenty eight (28) healthy subjects (21 males and 7 females) were enrolled in the study of which twenty seven (27) subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. All volunteers selected for this study will be healthy men or women 18 years of age or older at the time of dosing.
2. The weight range will not exceed ± 20 % for height and body frame as per desirable weights for adult - 1983 Metropolitan Height and Weight Table
3. If female and:

Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator (s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or Is postmenopausal for at least 1 year; or Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

1. Volunteers with a recent history of drug or alcohol addiction or abuse
2. Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system (s) or psychiatric disease (as determined by the clinical investigators)
3. Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
4. Volunteers demonstrated a positive hepatitis B surface antigen screen or a reactive HIV antibody screen
5. Volunteers demonstrating a positive drug abuse screen when screened for this study
6. Female volunteers demonstrating a positive pregnancy screen
7. Female volunteers who are currently breast feeding
8. Volunteers with history of allergic response(s) to Gabapentin or related drugs
9. Volunteers with a history of clinically significant allergies including drug allergies
10. Volunteers with a history of clinically significant illness during the 4 weeks prior to period I dosing (as determined by the clinical investigators)
11. Volunteers who currently use tobacco products
12. Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to period I dosing
13. Volunteers who report donating greater than 150 mL of the blood within 30 days prior to period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
14. Volunteers who have donated plasma (eg. Plasmapheresis) within 14 days prior to period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
15. Volunteers who report receiving any investigational drug within 30 days prior to period I dosing
16. Volunteers who report taking any systemic prescription medication in the 14 days prior to period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-10; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html